CLINICAL TRIAL: NCT02403596
Title: Study ESPER: Blood-sparing During the Placement of a Total Hip Prosthesis With the Exacyl® in Patients Treated With Rivaroxaban, Phase IV
Brief Title: Blood-sparing During Hip Prosthesis Surgery With Exacyl® in Patients Treated With Rivaroxaban
Acronym: ESPER
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University Hospital, Brest (Other)
Collaborators: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ESPER; RB15.005 (Other: Brest UH)
Record Dates: First submitted 2015-03-13; First posted 2015-03-31 (Estimated); Last update posted 2018-01-09 (Actual); Status verified 2018-01

CONDITIONS: Blood Loss After a Total Hip Replacement
Keywords: Hip replacement; rivaroxaban; exacyl; blood loss
MeSH Terms: conditions — Hemorrhage | interventions — Tranexamic Acid

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Group 1: Exacyl®: Standard treatment (Experimental): Intravenous use. 1g Exacyl® at H0 (Hour = 0 in other term at the time of incision) then 1g Exacyl® at H+3 then 1g Exacyl® placebo at H+7 and H+11
  Interventions: Drug: Exacyl®; Other: Placebo of Exacyl®
- Group 2: Exacyl®: Extended treatment (Experimental): Intravenous use. 1g Exacyl® at H0 (Hour = 0 in other term at the time of incision) then 1g Exacyl® at H+3 / H+7 and H+11
  Interventions: Drug: Exacyl®
- Group 3: Placebo (Placebo Comparator): This group will receive a placebo of Exacyl®: 1g placebo of Exacyl® at H0 (Hour = 0 in other term at the time of incision) then 1g placebo of Exacyl® at H+3 / H+7 and H+11
  Interventions: Other: Placebo of Exacyl®

INTERVENTIONS:
Drug: Exacyl®
  Other Names: Tranexamic acid
  Arms: Group 1: Exacyl®: Standard treatment; Group 2: Exacyl®: Extended treatment
Other: Placebo of Exacyl®
  Arms: Group 1: Exacyl®: Standard treatment; Group 3: Placebo

SUMMARY:
This study evaluates the efficacy of tranexamic acid versus placebo on perioperative blood loss using two dosage regimens (standard and extended) after a surgery during total hip arthroplasty in patients receiving the novel fast-acting oral anticoagulant rivaroxaban for prophylaxis of thrombosis.

DETAILED DESCRIPTION:
In 2011, 140 000 total hip replacements were performed and bleeding remains one of the major complications responsible for significant morbidity. This study will evaluate a new treatment to prevent bleeding due to this surgery. Indeed, the tranexamic acid (Exacyl) will be used in two modes of administration (standard or extended) versus placebo combined with a Rivaroxaban treatment at a dose of 10 mg / day for 35 days.

Patients will be randomized (exacyl standard vs exacyl extended vs. placebo) and will be followed for 3 months.

ELIGIBILITY:
Inclusion Criteria:

* Over 18 years of age
* Scheduled to undergo elective non-traumatic primary cementless THA
* Having given written informed consent to participate in the trial
* Covered by Social Security

Exclusion Criteria:

* Rapidly destructive arthrosis of the hip
* History of prior surgery on the operative hip
* Contraindications to the use of tranexamic acid:

  * Ischaemic artery disease (angina pectoris, myocardial infarction, acute coronary syndrome or stroke)
  * History of venous thromboembolism
  * Severe renal impairment, i.e. with clearance < 30mL/mn
  * Epilepsy or history of convulsions
* Contraindications to the use of rivaroxaban

  * Severe renal failure (clearance <30ml / min)
  * Cirrhotic patients with Child Pugh B
  * Pregnancy and breastfeeding
* Cognitive disorder that precludes giving informed consent
* Refusal to participate in trial
* Allergy to either of the trial treatments
* On-going prophylaxis of thrombosis using an agent other than rivaroxaban
* On-going platelet aggregation inhibitor at a dose exceeding 125 mg daily

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 231 (Actual)
Dates: Start 2015-10-20 (Actual); Primary Completion 2017-08-29 (Actual); Study Completion 2017-08-29 (Actual)

PRIMARY OUTCOMES:
Total blood loss | Between Day-1of surgery and Day+3 of surgery (5 days)
  Total Blood Loss (TBL) in mL of red blood cells, calculated using Mercuriali's formula at 100% haematocrit (Ht) and then converted to mL of blood at 35% Ht

SECONDARY OUTCOMES:
Difference in haemoglobin level (g/dL) between Day-1 and Day+3 | 5 days
Maximum difference in haemoglobin level (g/dL) from D-1 up to D+3 | 5 days
Number of transfusions and volume in mL performed during hospitalisation (operating theatre and unit) | 5 days
Major haemorrhagic events, clinically significant non-major haemorrhagic events and minor haemorrhagic events | 3 month
Surgical revision | 3 month
Occurrence of venous or arterial thromboembolic events | 3 month
Local infectious complications | 3 month
Death due to any cause and death due to cardiovascular cause | 3 month

CONTACTS AND LOCATIONS:
Locations (4):
- France (4):
  - HIA Clermont Tonnerre Brest, Brest
  - Polyclinique de Keraudren, Brest
  - CHRU Brest, Brest
  - CH Morlaix, Morlaix